Effect of transversus abdominis plane block combined with general anesthesia on perioperative stress response in patients undergoing radical gastrectomy

NCT number: NCT03035916

2017.1.30

## Informed Consent Form

Effect of transversus abdominis plane block combined with general anesthesia on perioperative stress response in patients undergoing radical gastrectomy: A randomized controlled study.

| NAME: | No.: |
|-------|------|
| - | |

Transabdominal radical gastrectomy is an effective strategy for treatment of malignant gastric disease. However, the excessive stress and immunologic response induced by surgeries are to be a disadvantage of postoperative rehabilitation, especially among patients with systemic disease and malignant tumor. In order to improve the effect of postoperative analgesia, to enhance postoperative recovery, we are going to conduct a clinical study on postoperative analgesia and systemic stress response after gastrectomy (Subject number: 3D5l4L463430), the purpose of the study is to verify the effect of abdominal transverse

obstruction on reducing postoperative pain and the stress intensity of the body. All the clinical data obtained will be used for the treatment and scientific research.

Here we need to explain to you in the following:

- The treatment used in this study confirmed to be useful on the patient's perioperative recovery after a large number of basic and clinical studies. But as any other treatment, this one may produce some adverse reactions. Once there are some adverse reactions, we will take timely and effective measures to minimize the damage.
- 2. There will not be any additional medical expenses for participants in this study.
- 3. Only relevant doctors and researchers will know the patient's information. We will not provide this information to others without your permission.
- 4. Participation in the study is entirely voluntary, during the study you and your family have the right to withdraw from the study at any time. If the patient is not eligible for the study for some

special reason, the doctor has the right to terminate your participation in the study. We will do our best to provide standardized treatment and services. Hope you or your family will work with the doctors.

If you and your family decide to participate in this study, please read the statement carefully.

| I have read the statement and agreed to |
|-----------------------------------------|
| participate in this study. |
| Signature: |